CLINICAL TRIAL: NCT02456220
Title: Three-dimensional Assessment of the Dentoskeletal Changes Associated With Herbst Appliance Therapy: A Controlled Clinical Trial
Brief Title: Dentoskeletal Changes Associated With Herbst Appliance Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bernardo Quiroga Souki (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor-Investigator, Bernardo Quiroga Souki, PhD, Pontifícia Universidade Católica de Minas Gerais
Organization: Pontifícia Universidade Católica de Minas Gerais (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUCMinasGerais
Record Dates: First submitted 2015-05-25; First posted 2015-05-28 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Malocclusion, Angle Class II
Keywords: Herbst appliance; Computed tomography; 3D imaging; Growth and development; Orthodontic Appliances, Functional
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Orthodontic Appliances, Functional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Herbst Group (Experimental): Patients treated with Herbst appliance.
  Interventions: Device: Herbst appliance
- Comparison Group (No Intervention): Patients that received only teeth movement (alignment and leveling before Herbst insertion), without any orthopedic intervention.

INTERVENTIONS:
Device: Herbst appliance — Group treated with conventional Herbst appliance for mandibular advancement during orthopedic treatment.
  Arms: Herbst Group

SUMMARY:
The aim of the study is to perform a three-dimensional (3D) evaluation of the dentoskeletal changes in pubertal Class II malocclusion subjects treated with the Herbst appliance (HAG), in comparison with a Class II comparison group (CG). 3D virtual models generated from three time-point CBCTs (T0, baseline; T1, immediately after Herbst insertion; and T2, 8 months after) of 25 HAG patients will be evaluated. Virtual models obtained from 25 Class II malocclusion patients, in the same stage of biologic maturation and skeletal abnormality, but with no orthopedic treatment will be constructed for the CG subjects. These CG patients are under orthodontic treatment, but only with teeth alignment. Voxel based registration on the anterior cranial fossa will be used to assess maxillary and mandibular displacement/articular fossa remodeling; regional registration on the mandibular corpus will be performed to evaluate mandibular growth and mandibular dental changes; and regional registration on the anterior region of the maxilla will be performed to evaluate maxillary growth and maxillary dental changes.

DETAILED DESCRIPTION:
1. BACKGROUND Class II malocclusion is highly prevalent worldwide, and it is a major reason for orthodontic treatment to be initiated. This type of malocclusion can be restricted to the dentoalveolar region, but the majority of Class II patients exhibit a strong skeletal component to the malocclusion, including most frequently mandibular skeletal retrusion and an increased lower anterior facial height. With increased severity of the mandibular deficiency, the orthodontist is challenged to treat the underlying skeletal problem appropriately.

   For growing patients, the use of fixed and removable mandibular advancement appliances has been advocated for many decades. A variety of fixed Herbst appliance designs have achieved worldwide acceptance in that they eliminate most major patient compliance factors. Today the Herbst appliance (HA) is by far the most frequently used mandibular jumping device in the United States, with more Herbst appliance being fabricated than all other functions appliances combined.

   The Herbst appliance originally was introduced by Emil Herbst in the early years of the twentieth century, but it did not achieved worldwide clinical acceptance until its re-introduction by Hans Pancherz 70 years later. Since then, a significant number of clinical and scientific studies has been conducted about HA, particularly by Pancherz and colleagues.

   Two-dimensional cephalometric studies have reported increases in the length of the mandible and in forward displacement of the mandible following HA in comparison to matched untreated controls. On average, 2 mm of mandibular length gain (measured from Gonion to Pogonion) and 1.5 degree of improvement in the SNB angle can be observed following Herbst appliance therapy.

   Investigations in experimental animals have provided the histological evidence of the changes in the condyles, rami, and articular fossae when the mandible is advanced in a laboratory setting. Previous reports have showed an increased proliferation of the condylar cartilage in monkeys that had their mandible advanced with the Herbst appliance. These adaptations occurred primarily in the posterior and posterosuperior regions of the condyle. They also reported significant bone deposition along the posterior border of the mandibular ramus during the early part of the experimental period as well as significant deposition of new bone on the anterior surface of the postglenoid spine at the articular fossae. It should be noted, however, that the post-glenoid spine is not well-defined in humans.

   Clinical investigations using Magnetic Ressonance Imaging (MRI) and lateral radiographs have showed that changes in the mandibular condyles and articular fossae may occur with Herbst therapy. It has been demonstrated that following Herbst therapy some articular fossa remodeling can be seen at the anterior surface of the postglenoid spine, which causes a relocation of the articular fossae in a downward and forward direction. But such fossa adaptation in Herbst patients is less extensive than in experimental animals, with much individual variation in response evident.

   Although most Herbst studies are convergent as to the extent of skeletal and dentoalveolar adaptations, some questions still remain:
   * How much mandibular growth can be achieved with therapeutic mandibular advancement?
   * How much mandibular rotation and skeletal bite opening occurs?
   * How much of the original mandibular advancement is maintained long-term?
   * Is there is an adaptive behavior of the articular fossa after mandibular advancement, with bone remodeling occurring in the fossa.

   In the last decade, a new methodology using 3D virtual modeling has been developed allowing a change in the paradigm of assessing the skeletal changes associated with growth and treatment; this technology that has opened new horizons in scientific investigations of dentofacial orthopedics. Recently, the American Journal of Orthodontists and Dentofacial Orthopedics published the first 3D report on Herbst treatment, a pilot study in which 7 Class II subjects treated with the Herbst appliance were compared with 7 Class II subjects treated with fixed appliances and intermaxillary elastics. It was reported that Class II patients undergoing Herbst treatment demonstrated anterior displacement of the condyles and articular fossae along with maxillary restraint when compared with the Class II patients used for comparison.

   The aim of the present prospective controlled clinical trial is to investigate the skeletal changes in the mandible and articular fossae in Class II patients undergoing Herbst appliance therapy, using 3D virtual models in comparison to a control group comprising Class II subjects.
2. PATIENTS AND METHODS b.1) Study design

This is a non-randomised controlled clinical trial, with intervention. Two groups are been planned: 1) Class II malocclusion subjects treated with Herbst appliance (HAG); and 2) Class II malocclusion subjects treated only with teeth alignment. The two groups are matched by stage of skeletal maturation, type of malocclusion, chronological age, and gender. There is no blinding for the outcome evaluators. Due to ethical concerns, the comparison group will be composed of Class II subjects that need previous alignment and leveling of the teeth before orthopedic phase of their treatment.

b.2) Participants - settings and location where the data are collected The treatment are been performed in the Orthodontic Clinic of Pontifical Catholic University of Minas Gerais (Belo Horizonte, Brazil). This is a private university, but the patients are mostly low-income subjects. Data has been collected from August 2013 and finished on September 2015.

b3) Sample size Based on the standard deviation of 1.85 mm reported by Pancherz et al.28, an alpha significance level of 0.05 and a power of 0.80 to detect changes of 1.5 mm, a preliminary sample size of 25 patients per group was calculated.

Therefore, 25 individuals have received a Herbst appliance at the beginning of their treatment with a one-step full activation - Herbst Appliance Group (HAG); while 25 skeletal Class II malocclusion individuals, with indication for HA therapy, but with other clinical conditions that required prior treatment before HA insertion, have been allocated to the CG. The two groups have been matched by chronological age (between 12 years and 16 years-old), by stage of skeletal maturation and by the stage of dental development (permanent dentition).

b4) Appliance design

The Herbst appliance design included bilateral telescoping arms (3M Abzil, São José do Rio Preto, Brazil) articulated with pivots that were positioned in both the maxillary and mandibular arches. The pivots were welded to a rigid cantilever wire (.040-in stainless steel) extending from the lower first permanent molar bands (TP Orthodontics, La Porte, IN) to the canine regions of the mandible. In the maxillary arch, the pivots were welded to bands on the permanent first molars. A Hyrax expander (Morelli Ortodontia, Sorocaba, Brazil) and a .040-in stainless steel (SS) lower lingual arch were added to the HA structure to improve appliance stability and transverse dimensional control. Two .028-in SS wires were used as occlusal rests in the permanent second molars to avoid their extrusion after activation. The occlusal rests were removed when they interfered with the occlusion to avoid bite opening.

b5) Method of registration

Cone beam computed tomography (CBCT), intra-oral pictures, and extra-oral pictures have been collected in three time-points for HAG (T0, T1, and T2), and in two time-point for CG (T0, and T2), as a regular protocol of orthodontic record for these clinical treatments.

b6) Method of measurement

Analysis of serial CBCT images to evaluate changes between T0, T1, and T2 include 3D analysis methodology using ITK-SNAP (open-source software, www.itksnap.org); SLICER (open-source software, www.slicer.org; and VAM - Vectra Analysis Model software version 3.7.6 (Canfield Scientific Inc., Fairfield, NJ). The tridimensional image analysis procedures included: (1) approximation of scans; (2) construction of 3D label models; (3) voxel based image registration; and (4) quantitative and qualitative assessments using 3D mesh surface models.

Quantitative assessment of the positional changes between the 3D surface models of the cranial base, maxilla, and mandible will be performed using point-to-point landmarks measurements (VAM software), and virtual analytics (SLICER software).

Interactive visual analytics include graphic displays with qualitative assessments using semitransparent overlays of the 3D surface models at the different time-points and quantitative assessments of the surface displacements using color-coded surface distance maps. All visual analytics assessments will be performed using two modules (Model-to-Model Distance and Shape Population Viewer) in the SLICER software.

Voxel based registration on the anterior cranial fossae will be used to assess maxillary and mandibular displacement/articular fossae remodeling; regional registration on the mandibular symphysis will be performed to evaluate mandibular growth and mandibular dental changes; and regional registration on the anterior region of the maxilla will be performed to evaluate maxillary growth and maxillary dental changes.

b7) Method of analysis

For the primary and secondary outcome measures it will be used Statistical Package for the Social Science (SPSS) software (version 16.0 Chicago, IL). Descriptive statistics will be presented for both groups. Statistical differences between the two groups will be calculated with Mann-Whitney test (comparison between the difference of the means of the HAG and CG). The comparison between the changes within each group will be performed using the Wilcoxon's test.

ELIGIBILITY:
Inclusion Criteria:

* Class II malocclusion with mandibular retrognathism
* Convex Profile
* Pubertal period
* Permanent dentition
* Parental permission with a signed consent form

Exclusion Criteria:

* Syndromic patients
* Previous orthopedic treatment

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Skeletal mandibular growth after Herbst appliance therapy | 8 months
  To test the mandibular rotation immediately after Herbst appliance insertion; and 2) to compare the displacement of the condyles with the reduction of overjet (OJ) and overbite (OB). Virtual 3D surface models of 25 subjects were generated from the cone-beam computed tomographs taken before treatment, and immediately after Herbst installation. Scans were registered on the cranial bases, and analyzed using point-to-point measurements, color-coded maps and semitransparent overlays.

SECONDARY OUTCOMES:
Mandibular displacement after Herbst appliance therapy | 8 months
  Based on cranial base volumetric superimposition, the assessment of the mandibular displacement will be performed. Based on regional superimposition of the mandibular corpus, the condilar and ramus growth will be evaluated.
Displacement of the mandibular condyles immediately after Herbst appliance insertion - 3D assessment | 5 weeks
  To test the mandibular rotation immediately after Herbst appliance insertion; and 2) to compare the displacement of the condyles with the reduction of overjet (OJ) and overbite (OB). Virtual 3D surface models of 25 subjects were generated from the cone-beam computed tomographs taken before treatment, and immediately after Herbst installation. Scans were registered on the cranial bases, and analyzed using point-to-point measurements, color-coded maps and semitransparent overlays.Scans were registered on the cranial bases, and analyzed using point-to-point measurements, color-coded maps and semitransparent overlays.
Maxillary displacement after Herbst appliance therapy | 8 months
  Evaluation of the maxillary displacement at the end of the treatment with the reference of the cranial base.
Bone remodeling of the articular fossae after Herbst appliance therapy | 8 months
  Evaluation of the bone remodeling of the articular fossae at the end of the treatment with the reference of the cranial base.
Dental positional changes after Herbst appliance therapy | 8 months
  Evaluation of the teeth movement at the end of the treatment with the reference of the maxilla and the mandible.

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Q Souki, PhD, Principal Investigator — Pontifícia Universidade Católica de Minas Gerais; James A McNamara Jr., PhD, Study Director — University of Michigan; Lucia Helena S Cevidanes, PhD, Study Chair — University of Michigan
Locations (1):
- Pontifícia Universidade Católica de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Buschang PH, Tanguay R, Demirjian A, LaPalme L, Turkewicz J. Mathematical models of longitudinal mandibular growth for children with normal and untreated Class II, division 1 malocclusion. Eur J Orthod. 1988 Aug;10(3):227-34. doi: 10.1093/ejo/10.3.227. No abstract available. PMID 3181302
- [Background] Buschang PH, Martins J. Childhood and adolescent changes of skeletal relationships. Angle Orthod. 1998 Jun;68(3):199-206; discussion 207-8. doi: 10.1043/0003-3219(1998)0682.3.CO;2. PMID 9622756
- [Background] Cevidanes LH, Oliveira AE, Grauer D, Styner M, Proffit WR. Clinical application of 3D imaging for assessment of treatment outcomes. Semin Orthod. 2011 Mar 1;17(1):72-80. doi: 10.1053/j.sodo.2010.08.012. PMID 21516170
- [Background] Cevidanes LH, Heymann G, Cornelis MA, DeClerck HJ, Tulloch JF. Superimposition of 3-dimensional cone-beam computed tomography models of growing patients. Am J Orthod Dentofacial Orthop. 2009 Jul;136(1):94-9. doi: 10.1016/j.ajodo.2009.01.018. PMID 19577154
- [Background] Hagg U, Rabie AB, Bendeus M, Wong RW, Wey MC, Du X, Peng J. Condylar growth and mandibular positioning with stepwise vs maximum advancement. Am J Orthod Dentofacial Orthop. 2008 Oct;134(4):525-36. doi: 10.1016/j.ajodo.2006.09.064. PMID 18929270
- [Background] Hagg U, Pancherz H. Dentofacial orthopaedics in relation to chronological age, growth period and skeletal development. An analysis of 72 male patients with Class II division 1 malocclusion treated with the Herbst appliance. Eur J Orthod. 1988 Aug;10(3):169-76. doi: 10.1093/ejo/10.3.169. No abstract available. PMID 3181295
- [Background] Kinzinger G, Kober C, Diedrich P. Topography and morphology of the mandibular condyle during fixed functional orthopedic treatment --a magnetic resonance imaging study. J Orofac Orthop. 2007 Mar;68(2):124-47. doi: 10.1007/s00056-007-0650-0. English, German. PMID 17372710
- [Background] LeCornu M, Cevidanes LH, Zhu H, Wu CD, Larson B, Nguyen T. Three-dimensional treatment outcomes in Class II patients treated with the Herbst appliance: a pilot study. Am J Orthod Dentofacial Orthop. 2013 Dec;144(6):818-30. doi: 10.1016/j.ajodo.2013.07.014. PMID 24286905
- [Background] Pancherz H, Malmgren O, Hagg U, Omblus J, Hansen K. Class II correction in Herbst and Bass therapy. Eur J Orthod. 1989 Feb;11(1):17-30. doi: 10.1093/oxfordjournals.ejo.a035960. PMID 2714389
- [Background] Pancherz H. The effect of continuous bite jumping on the dentofacial complex: a follow-up study after Herbst appliance treatment of class II malocclusions. Eur J Orthod. 1981;3(1):49-60. doi: 10.1093/ejo/3.1.49. No abstract available. PMID 6939593
- [Background] Pancherz H. The mechanism of Class II correction in Herbst appliance treatment. A cephalometric investigation. Am J Orthod. 1982 Aug;82(2):104-13. doi: 10.1016/0002-9416(82)90489-4. PMID 6961781
- [Background] Pancherz H. Vertical dentofacial changes during Herbst appliance treatment. A cephalometric investigation. Swed Dent J Suppl. 1982;15:189-96. PMID 6963773
- [Background] Pancherz H. The Herbst appliance--its biologic effects and clinical use. Am J Orthod. 1985 Jan;87(1):1-20. doi: 10.1016/0002-9416(85)90169-1. PMID 3855346
- [Background] Pancherz H. The nature of Class II relapse after Herbst appliance treatment: a cephalometric long-term investigation. Am J Orthod Dentofacial Orthop. 1991 Sep;100(3):220-33. doi: 10.1016/0889-5406(91)70059-6. PMID 1877546
- [Background] Pancherz H, Anehus-Pancherz M. Muscle activity in class II, division 1 malocclusions treated by bite jumping with the Herbst appliance. An electromyographic study. Am J Orthod. 1980 Sep;78(3):321-9. doi: 10.1016/0002-9416(80)90277-8. No abstract available. PMID 6931496
- [Background] Pancherz H, Fackel U. The skeletofacial growth pattern pre- and post-dentofacial orthopaedics. A long-term study of Class II malocclusions treated with the Herbst appliance. Eur J Orthod. 1990 May;12(2):209-18. doi: 10.1093/ejo/12.2.209. PMID 2351206
- [Background] Pancherz H, Fischer S. Amount and direction of temporomandibular joint growth changes in Herbst treatment: a cephalometric long-term investigation. Angle Orthod. 2003 Oct;73(5):493-501. doi: 10.1043/0003-3219(2003)0732.0.CO;2. PMID 14580015
- [Background] Pancherz H, Hagg U. Dentofacial orthopedics in relation to somatic maturation. An analysis of 70 consecutive cases treated with the Herbst appliance. Am J Orthod. 1985 Oct;88(4):273-87. doi: 10.1016/0002-9416(85)90126-5. PMID 3863486
- [Background] Pancherz H, Hansen K. Mandibular anchorage in Herbst treatment. Eur J Orthod. 1988 May;10(2):149-64. doi: 10.1093/ejo/10.2.149. No abstract available. PMID 3164681
- [Background] Pancherz H, Hansen K. Occlusal changes during and after Herbst treatment: a cephalometric investigation. Eur J Orthod. 1986 Nov;8(4):215-28. doi: 10.1093/ejo/8.4.215. No abstract available. PMID 3466794
- [Background] Pancherz H, Ruf S, Kohlhas P. "Effective condylar growth" and chin position changes in Herbst treatment: a cephalometric roentgenographic long-term study. Am J Orthod Dentofacial Orthop. 1998 Oct;114(4):437-46. doi: 10.1016/s0889-5406(98)70190-8. PMID 9790329
- [Background] Rabie AB, Tsai MJ, Hagg U, Du X, Chou BW. The correlation of replicating cells and osteogenesis in the condyle during stepwise advancement. Angle Orthod. 2003 Aug;73(4):457-65. doi: 10.1043/0003-3219(2003)0732.0.CO;2. PMID 12940568
- [Background] Ruf S, Pancherz H. Temporomandibular joint growth adaptation in Herbst treatment: a prospective magnetic resonance imaging and cephalometric roentgenographic study. Eur J Orthod. 1998 Aug;20(4):375-88. doi: 10.1093/ejo/20.4.375. PMID 9753819
- [Background] Ruf S, Pancherz H. Temporomandibular joint remodeling in adolescents and young adults during Herbst treatment: A prospective longitudinal magnetic resonance imaging and cephalometric radiographic investigation. Am J Orthod Dentofacial Orthop. 1999 Jun;115(6):607-18. doi: 10.1016/s0889-5406(99)70285-4. PMID 10358242
- [Background] Ruf S, Pancherz H. Herbst/multibracket appliance treatment of Class II division 1 malocclusions in early and late adulthood. a prospective cephalometric study of consecutively treated subjects. Eur J Orthod. 2006 Aug;28(4):352-60. doi: 10.1093/ejo/cji116. Epub 2006 Apr 27. PMID 16644850
- [Background] Ruf S, Wusten B, Pancherz H. Temporomandibular joint effects of activator treatment: a prospective longitudinal magnetic resonance imaging and clinical study. Angle Orthod. 2002 Dec;72(6):527-40. doi: 10.1043/0003-3219(2002)0722.0.CO;2. PMID 12518944
- [Background] Serbesis-Tsarudis C, Pancherz H. "Effective" TMJ and chin position changes in Class II treatment. Angle Orthod. 2008 Sep;78(5):813-8. doi: 10.2319/082707-391.1. PMID 18298212
- [Background] Voudouris JC, Woodside DG, Altuna G, Kuftinec MM, Angelopoulos G, Bourque PJ. Condyle-fossa modifications and muscle interactions during herbst treatment, part 1. New technological methods. Am J Orthod Dentofacial Orthop. 2003 Jun;123(6):604-13. doi: 10.1016/s0889-5406(03)00149-5. PMID 12806337
- [Background] Voudouris JC, Woodside DG, Altuna G, Angelopoulos G, Bourque PJ, Lacouture CY, Kuftinec MM. Condyle-fossa modifications and muscle interactions during Herbst treatment, Part 2. Results and conclusions. Am J Orthod Dentofacial Orthop. 2003 Jul;124(1):13-29. doi: 10.1016/s0889-5406(03)00150-1. PMID 12867894
- [Background] Woodside DG, Metaxas A, Altuna G. The influence of functional appliance therapy on glenoid fossa remodeling. Am J Orthod Dentofacial Orthop. 1987 Sep;92(3):181-98. doi: 10.1016/0889-5406(87)90411-2. PMID 3477085